CLINICAL TRIAL: NCT02089737
Title: Vectibix for Intravenous Infusion 100 mg and 400 mg Special Drug Use Surveillance "Survey on Unresectable, Advanced or Recurrent Colorectal Cancer With Wild-type KRAS Gene" (All-patient Surveillance)
Brief Title: Panitumumab for Intravenous Infusion 100 mg and 400 mg Special Drug Use Surveillance "Survey on Unresectable, Advanced or Recurrent Colorectal Cancer With Wild-type KRAS Gene" (All-patient Surveillance)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 183-011; JapicCTI-132374 (Registry Identifier: JapicCTI); JapicCTI-R140654 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-03-13; First posted 2014-03-18 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Advanced or Recurrent Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Panitumumab 6 mg/kg: Panitumumab 6 mg/kg, intravenous drip infusion over a 60-minute period, once every 2 weeks
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Panitumumab for intravenous infusion
  Other Names: Vectibix

SUMMARY:
The efficacy and safety of panitumumab (Vectibix) in the routine clinical setting will be studied.

Specifically, information will be collected on the following as events of interest: skin disorders, interstitial lung disease, infusion reactions, electrolyte abnormalities, and cardiac disorders.

DETAILED DESCRIPTION:
The efficacy and safety of panitumumab (Vectibix) in the routine clinical setting will be studied.

Participants of this surveillance will be patients with unresectable, advanced or recurrent colorectal cancer with the wild-type KRAS gene. The planned sample size is 2,000 patients.

The usual adult dosage is 6 mg/kg of panitumumab given by intravenous drip infusion over a 60-minute period once every 2 weeks. The dosage may also be reduced as needed, depending on the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, advanced or recurrent colorectal cancer with wild-type KRAS gene

Exclusion Criteria:

* Patients with a medical history of severe hypersensitivity to any of the ingredients of Vectibix

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unresectable, advanced or recurrent colorectal cancer with wild-type KRAS gene
Sampling Method: Non-Probability Sample
Enrollment: 3091 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled during the period from June 1, 2010 to November 14, 2010 were surveyed.
Pre-assignment Details: Surveyed participants had a clinical diagnosis of wild-type KRAS unresectable advanced/recurrent colorectal cancer.
Groups:
- Panitumumab: Panitumumab 6 mg/kg, intravenous drip infusion over a 60-minute period, once every 2 weeks for up to 42 weeks
Period: Overall Study
Arm/Group | Panitumumab
Started | 3091
Completed | 3085
Not Completed | 6
Not completed — Survey form not completed | 5
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Population: 3086 participants completed the survey form (5 participants did not complete it). 3085 participants were included in the safety analysis set after excluding 1 participant due to missing panitumumab treatment and AE data. From that set, 3084 participants were included in the efficacy analysis set after excluding 1 participant with missing data.
Arm/Group | Panitumumab
Number analyzed (Participants) | 3085
Age, Customized [Number; unit: Participants]
  < 75 years | 2582
  >= 75 years | 503
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1120
  Male | 1965
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3085
Region of Enrollment [Number; unit: Participants]
  Japan | 3085
KRAS genotype [Number; unit: Participants]
  Wild type | 3003
  Non-measurable/non-assessable | 78
  Mutant | 3
  Not determined | 1
  Unknown | 0
Treatment stage (excluding posteroperative adjuvant chemotherapy) [Number; unit: Participants]
  First-line | 310
  Second-line | 543
  Third-line or later | 2232
  Unknown | 0
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) at baseline [Number; unit: Participants] — ECOG-PS is measured on 6-point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all selfcare, but unable to carry out any work activities; 3=Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4=Completely disabled, cannot carry on any selfcare, totally confined to bed or chair; 5=Dead.
  Participants
    PS:0 | 1877
    PS:1 | 942
    PS:2 | 241
    PS:3 | 22
    PS:4 | 3
    Unknown | 0
Metastatic lesions/sites of relapse [Number; unit: Participants]
  No | 38
  Yes | 3046
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: The number of participants with adverse drug reactions reported during the observation period were tabulated by type, seriousness, and time of onset. . Adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug to the last dose of study drug.
Time Frame: Baseline through Week 42
Population: Of the 3086 participants who completed the survey form, 3085 participants were included in the safety analysis set after excluding 1 participant for whom information regarding panitumumab treatment and adverse events were missing.
Measure: Number; unit: Participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 3085
Participants
  Frequency of adverse drug reactions | 2595
  MedDRA SOC: Skin and subcutaneous tissue disorders | 2364
  MedDRA SOC: Infections and infestations | 771
  MedDRA SOC: Gastrointestinal disorders | 642
  MedDRA SOC: Metabolism and nutrition disorders | 552
  MedDRA SOC: Cardiac disorders | 7

2. Secondary Outcome: Progression-free Survival
Description: Progression-free Survival (PFS) was defined as the time from the first day of study treatment to documented disease progression or death on study. For participants who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: Up to Week 42 or death (whichever occurred first)
Population: Participants who were included in the efficacy analysis set and received panitumumab monotherapy as a third-line or later therapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab
Number analyzed (Participants) | 1061
Months | 3.5 [3.3 to 4.0]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time to death from the start of panitumumab administration was tabulated.
Time Frame: Up to Week 42 or death (whichever occurred first)
Population: All participants that received panitumumab monotherapy as a third-line or later therapy.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 1061
weeks | 41 [36 to 47]

ADVERSE EVENTS:
Time Frame: For up to 42 weeks
Description: Serious adverse events were tabulated dividing into 2 groups: panitumumab monotherapy or concomitant administration of panitumumab and chemotherapy Serious adverse events grouped by organ system, with number and frequency of such events.
Arm/Group | Panitumumab | Concomitant Administration of Panitumumab and Chemotherapy
Serious Adverse Events (participants affected / at risk) | 614/1254 | 747/1831
Other Adverse Events (participants affected / at risk) | 640/1254 | 1084/1831
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=1254) | Concomitant Administration of Panitumumab and Chemotherapy (N=1831)
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1
Endocarditis (Infections and infestations) | 0 | 1
Fungaemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Liver Abscess (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Necrotizing fasciitis (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 3 | 5
Pneumonia (Infections and infestations) | 2 | 12
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 6
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 5 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Device-related infection (Infections and infestations) | 1 | 2
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Infectious peritonitis (Infections and infestations) | 1 | 1
Bile duct cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 524 | 557
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 17
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 10
Tetany (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 16
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 1
Bulbar palsy (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 5 | 3
Convulsion (Nervous system disorders) | 2 | 4
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 2
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Peripheral neuropathy (Nervous system disorders) | 0 | 1
Paralysis (Nervous system disorders) | 1 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 2
Periorbital oedema (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Unstable angina (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung diseases (Respiratory, thoracic and mediastinal disorders) | 16 | 27
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 26
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 3 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 6 | 7
Intestinal obstruction (Gastrointestinal disorders) | 5 | 6
Malaena (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 5
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal performation (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 24
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 5
Subileus (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Oral mucosa erosion (Gastrointestinal disorders) | 1 | 0
Ileal fistula (Gastrointestinal disorders) | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 3
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 4
Jaundice (Hepatobiliary disorders) | 0 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 14
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Oculomucocutaneous syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 4
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 3 | 1
Chills (General disorders) | 1 | 0
Death (General disorders) | 3 | 4
Fatigue (General disorders) | 2 | 2
Gait disturbance (General disorders) | 1 | 0
Malaise (General disorders) | 4 | 10
Multi-organ failure (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 7
Device occlusion (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood calcium decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 13
Platelet count descreased (Investigations) | 2 | 3
White blood cell count decreased (Investigations) | 1 | 10
White blood cell count increased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 3
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 12
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=1254) | Concomitant Administration of Panitumumab and Chemotherapy (N=1831)
Paronychia (Infections and infestations) | 269 | 458
Hypomagnesaemia (Metabolism and nutrition disorders) | 218 | 198
Diarrhoea (Gastrointestinal disorders) | 30 | 155
Stomatitis (Gastrointestinal disorders) | 123 | 463
Acne (Skin and subcutaneous tissue disorders) | 81 | 112
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 617 | 959
Dry skin (Skin and subcutaneous tissue disorders) | 265 | 344
Rash (Skin and subcutaneous tissue disorders) | 98 | 160

LIMITATIONS AND CAVEATS:
The present specified drug-use survey is a one-arm observational study with no control group. Therefore, the observed outcome measures provide exploratory information regarding these endpoints; however, do not constitute verification results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.